CLINICAL TRIAL: NCT06179537
Title: A Phase I, Double-Blind, Randomised, Adaptive-designed Study to Assess the Pharmacokinetics and Safety of BLU-5937 in Healthy Adult Japanese and Caucasian Subjects Following Single and Multiple Oral Doses
Brief Title: Evaluation of the Pharmacokinetics and Safety of BLU-5937 in Healthy Adult Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUS-P1-07
Record Dates: First submitted 2023-11-27; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — BLU-5937

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 10 Japanese and 8 Caucasian subjects. 8 out of 10 Japanese subjects will receive BLU-5937 Dose A and 2 will receive placebo. All Caucasian subjects will receive BLU-5937 Dose A.
  Interventions: Drug: BLU-5937
- Cohort 2 (Experimental): 8 Japanese subjects. 6 out of 8 will receive BLU-5937 Dose B and 2 will receive placebo.
  Interventions: Drug: BLU-5937
- Cohort 3 (Experimental): 8 Japanese subjects. 6 out of 8 will receive BLU-5937 Dose C and 2 will receive placebo.
  Interventions: Drug: BLU-5937

INTERVENTIONS:
Drug: BLU-5937 — Single and multiple doses assessment

SUMMARY:
This is a Phase I, Double-Blind, Randomised, Adaptive-designed Study to Assess the Pharmacokinetics and Safety of BLU-5937 in Healthy Adult Japanese and Caucasian Subjects Following Single and Multiple Oral Doses

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females

Exclusion Criteria:

* History of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Assessment of ECG QTcF interval (ms) change | Pre-dose up to 48 hours post-dose for both single and multiple administration
Assessment of diastolic and systolic blood pressure (mmHg) change | Pre-dose up to 48 hours post-dose for both single and multiple administration
Assessment of heart rate (BPM) change | Pre-dose up to 48 hours post-dose for both single and multiple administration
Number of participants with clinically significant changes in Clinical laboratory tests | Pre-dose up to 48 hours post-dose for both single and multiple administration
Number of participants with clinically significant changes in Physical Examination | Pre-dose up to 48 hours post-dose for both single and multiple administration
Adverse Event and Adverse Event of medical interest monitoring | Pre-dose up to 48 hours post-dose for both single and multiple administration and again at follow-up call (1 week after discharge)
Measurement of the area under the plasma concentration by time curve (AUC) | Pre-dose up to 48 hours post-dose for both single and multiple administration
Measurement of the maximum observed plasma drug concentration (Cmax) | Pre-dose up to 48 hours post-dose for both single and multiple administration

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No